CLINICAL TRIAL: NCT03343522
Title: The Effects of Exercise Training in Vascular Function of Patients Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia de Laranjeiras (Other)
Collaborators: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Juliana Pereira Borges, Principal Investigator, Instituto Nacional de Cardiologia de Laranjeiras
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CAAE42162815.5.0000.5272
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: HIV/AIDS
Keywords: Vascular function; Physical training; Laser Speckle Contrast Imaging
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedentarism (No Intervention): Patients assigned to this arm shall not perform regular exercise training.
- Exercise Training (Experimental): Patients assigned to this arm will be enrolled in exercise training program.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — A multimodal exercise training program (aerobic, strength and flexibility exercises) for 6 months (60-min sessions performed 3 times/week with moderate intensity).
  Arms: Exercise Training

SUMMARY:
Introduction: It is well known that the infection caused by the Human Immunodeficiency Virus (HIV) is associated to a higher cardiovascular event risk. On the other hand, it is clear that the aerobic exercise training induces improvements in autonomic control and vascular function, through increases in vasodilator agents and blood vessels number. However, the investigators could not find previous works that studied the microvascular function in response to exercise training in HIV patients.

Objectives: To study the impact of aerobic exercise training in endothelial function of HIV patients. In addition, the investigators will verify the association of the physical fitness to the nitric oxide bioavailability, angiogenesis and lipid profile in HIV patients.

Methods: The study subjects will be composed by HIV patients, that will be randomly divided in two different groups: exercised and sedentary. The subjects will be tested before and after training in regards to endothelial function, nitric oxide bioavailability, physical fitness and lipid profile, through flowmetry, colorimetric essays, maximal cardiopulmonary exercise test, and biochemical tests; respectively. The exercise training will be performed in a treadmill for 12 weeks, 3 times a week, 40 minutes each section.

Expected Results: The investigators expect to achieve markers that will help in understanding the interaction of HIV with several factors that contribute to an increased endothelial function after exercise training.

DETAILED DESCRIPTION:
HIV-infection triggers a massive oxygen reactive species production, increasing oxidative stress and vascular complications. Despite the importance of therapeutic strategies in reducing the cardiovascular risk among HIV-infected patients (HIVP), exercise-related effects upon macro-and-microvascular endothelial function and oxidative stress in HIVP have not been previously reported.

ELIGIBILITY:
Inclusion Criteria:

* sedentarism for at least 6 months;
* diagnosis of HIV infection.

Exclusion Criteria:

* opportunistic diseases;
* nephropathies;
* cardiovascular diseases;
* locomotor limitations;
* liver diseases.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Skin microvascular blood flow | Baseline and 3 months
  Microvascular reactivity will be evaluated by laser speckle contrast imaging with laser wavelength of 785 nm in combination with iontophoresis of acetylcholine (ACh) and sodium nitroprusside (SNP) for noninvasive and continuous measurements of cutaneous microvascular flow changes in the forearm.

SECONDARY OUTCOMES:
Peak Oxygen consumption | Baseline and 3 months
  Measured at a maximal graded exercise test.
Nitrite/nitrate | Baseline and 3 months
  Colorimetric assay kit
Body fat | Baseline and 3 months
  Dual-energy X-ray absorptiometry.
Forearm macrovascular blood flow | Baseline and 3 months
  Forearm macrovascular blood flow will be evaluated by venous occlusion plethysmography.
Capillary density | Baseline and 3 months
  Capillary density will be evaluated by high-resolution intra-vital color microscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana P Borges, PhD, Principal Investigator — Insituto Nacional de Cardiologia and Rio de Janeiro State University
Locations (1):
- Rio de Janeiro State University, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No